CLINICAL TRIAL: NCT06243822
Title: Hemodynamic Effects of Ketamine Compared With Propofol as Continuous ICU Sedation in Mechanically Ventilated Patients
Brief Title: Ketamine Versus Propofol as ICU Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, mostafa saieed fahim mansour, lecturer of anaesthesiology, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1/2023ANET9
Record Dates: First submitted 2024-01-14; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Ketamine; Propofol; Sedation; Mechanical Ventilation
MeSH Terms: interventions — Ketamine; Propofol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine group (Active Comparator)
  Interventions: Drug: Ketamine
- propofol group (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ketamine — ketamine is initiated at 0.5 mg/kg/h and titrated by 0.25 mg/kg/h every 15 minutes to a maximum dosage of 4 mg/kg/h to achieve appropriate sedation.
  Arms: Ketamine group
Drug: Propofol — Propofol is initiated at 0.3 to 0.6 mg /kg/hr. and titrated by 0.3 to 0.6 mg/kg/h every 5 to 10 minutes up to a maximum dosage of 4.5 to 4.8 mg/kg/hr. to achieve appropriate sedation.
  Arms: propofol group

SUMMARY:
this study is to assess the hemodynamic profile of ketamine compared with propofol in critically ill, mechanically ventilated adult Patients study will be carried out on 100 mechanically ventilated patients who received one sedative agent propofol or ketamine The patients will be randomized into two equal groups to receive either ketamine or propofol Group 1 (Ketamine group): ketamine is initiated at 0.5 mg/kg/h and titrated by 0.25 mg/kg/h every 15 minutes to a maximum dosage of 4 mg/kg/h to achieve appropriate sedation. Group 2 (Propofol group): Propofol is initiated at 0.3 to 0.6 mg /kg/hr. and titrated by 0.3 to 0.6 mg/kg/h every 5 to 10 minutes up to a maximum dosage of 4.5 to 4.8 mg/kg/hr. to achieve appropriate sedation.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated, and receive sedation with continuous infusion propofol, or ketamine for at least 24 hours

Exclusion Criteria:

* Receiving propofol or ketamine concurrently.

  * Transferred from an outside hospital on sedation.
  * Receiving ketamine for an indication other than sedation.
  * Daily intake of opioids.
  * Contraindication to any drug used in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
heart rate | every 15 min for the first hour then every hour for next six hours then every six hours for 48 hours
  measure heart rate
mean arterial blood pressure | every 15 min for the first hour then every hour for next six hours then every six hours for 48 hours
  measure mean arterial blodd pressure

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Saieed Mansour, MD, Principal Investigator — Menoufia University
Locations (1):
- Menoufia University, Shibīn al Kawm, Menoufia, Egypt